CLINICAL TRIAL: NCT06012396
Title: Safety and Validation of Community Rehabilitation Exercise Program for Stroke Patients
Brief Title: Community-based Complex Exercise for Stroke Patients
Acronym: COB-CEPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sung-Hwa Ko, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNUYH_ETRI_3
Record Dates: First submitted 2023-08-06; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: rct
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: Stoke complex exercise program
- Daily life group (No Intervention)

INTERVENTIONS:
Behavioral: Stoke complex exercise program — 1. warm-up(5min) flexibility exercise - neck, triceps brachii, biceps brachii, forearm, back, quadriceps, biceps femoris, ankle
  2. main exercise(40min) aerobic exercise(20min)- use stepper, treadmill, high intensity HRR60%, RPE 11~14 low intensity HRR30%, RPE 9~11 repeated interval training strength and balance exercises(20min)- program1. upper(shoulder press, chest press, biceps curl), lower(hip flexion, knee extension), Core(plank exercise, sit up) program2. upper(seated back row, triceps extension), lower(hip extension, hip abduction, knee flexion, Core(superman exercise, bridge exercise) repeated ever other day program1, program2 clean-up(5min) - same as warm-up
  Arms: Exercise group

SUMMARY:
A lot of physical and social effects of exercise programs and daily physical education have already been proven for stroke patients after discharge. However, stroke patients have shown a passive attitude in participating in physical education or exercise programs for life, and the local community lacked appropriate guidelines or experience in guiding exercise and physical education for stroke patients, so they had a burden on instructing exercise. In this study, an appropriate complex exercise program was established for patients after discharge through analysis of domestic and foreign research data to provide an environment and opportunity to exercise in the community, and based on the results, stroke patients actively exercise in the community in the future. The goal is to provide a basis for doing so.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients aged 30 years or older residing in the community
* Those who can walk independently and have a score of 3 or higher in the Functional Ambulation Category (FAC)
* The daily life dependence of the stroke patient is a person who can perform simple tasks necessary for daily life, Those who scored 2 points or less on the Modified Rankin Scale (mRS)
* Subjects with no or mild stiffness of the affected upper and lower limbs, with a score of 1 or less on the Modified Ashworth Scale (MAS)
* All 3 major joints of the affected upper and lower limbs (Manual Muscle Test (MMT)) are 3 points (F grade) or higher ruler

Exclusion Criteria:

* With moderate or severe cognitive dysfunction, Korean-Mini Mental state test (Korean-Mini Mental state test) Those who scored less than 18 points in the Examination (K-MMSE)
* A person with a moderate or higher fall risk and less than 41 points on the Berg Balance Scale (BBS)
* Those who have difficulty understanding the intervention exercise program or expressing symptoms due to severe language impairment
* Those who cannot apply this intervention exercise program due to serious cardiovascular disease
* Those who have musculoskeletal disorders that make it impossible to exercise
* Those who are judged unsuitable for this study under the judgment of a specialist in rehabilitation medicine due to other diseases

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
6WMT | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  6-minute walk test practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians

SECONDARY OUTCOMES:
MRS | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability The scale runs from 0-6, running from perfect health without symptoms to death.
BBS | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Berg balance scale (0-56, the higher the better) Objectively determine a patient's ability to safely balance during a series of predetermined tasks
FAC | visit 1, visit 23
  Functional ambulation category (0-5, the higher the better) 6-point functional walking test that evaluates ambulation ability
MMT | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Manual Muscle Testing (MMT) is a technique used in physical therapy and rehabilitation to assess the strength and function of individual muscles or muscle groups. It involves the application of specific resistance against the muscle's movement to determine its ability to generate force.
  This technique includes assessing major muscles from the upper and lower limbs opposing the therapist's force and grading the patient's muscle strength on a 0 to 5 scale
TUG | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Timed up and go To determine fall risk and measure the progress of balance
Grip Strength | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Grip strength measure of muscular strength or the maximum force/tension generated by one's forearm muscles
Body composition | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Percentage of fat, bone, and muscle in the body
Physical activity | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  International Physical Activity Questionnaire (No scores) 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old
EQ-5D | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Euro-Quality of Life-5 Dimension (EQ-5D) (5-25, the higher the better) A brief and simple instrument measuring health related quality of life
GDS | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Getriatic depression scale (0-15, the higher the more depressive) Assessment of depression in the elderly
sit to stand | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Recording the number of times sitting and rising for 30 seconds by measuring the strength of the lower extremities of the elderly
flexibility test | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Measure the length beyond the tip of the toes with the hand stretched out in a seated forward bending position.
coordination test | Baseline and Follow-up evaluation (through study completion, an average of 6 weeks)
  Assessment of Coordination Measures in Older Adults. Draw a rectangle with a width of 3.6m and a length of 1.6m, place a chair at a point 2.4m from the center in both corners, and measure the time to return to the left and right rear corners twice in 0.1 second units

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided